CLINICAL TRIAL: NCT04657705
Title: Application of High Power Radio Frequency Energy in the Interventional Treatment of Patients With Ventricular Tachycardia and Structural Heart Disease
Brief Title: Application of High Power Radio Frequency Energy in the Ventricular Tachycardia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Collaborators: Meshalkin National Medical Research Center, Ministry of Health of Russian Federation (Other Government); Heart and Vascular Center Bad Bevensen, Germany (Unknown); National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government); National Research Center of Surgery, Russia (Other Government); I.M. Sechenov First Moscow State Medical University (Other); Texas Cardiac Arrhythmia Institute, Austin, Texas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BURN VT
Record Dates: First submitted 2020-09-18; First posted 2020-12-08 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Ventricular Tachycardia; Heart Diseases
Keywords: High Power Radio Frequency Energy; Ventricular Tachycardia; Structural Heart Disease
MeSH Terms: conditions — Tachycardia, Ventricular; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High power ablation (Experimental): High power ablation parameters (50-55 W)
  Interventions: Procedure: High power ablation
- Standard ablation power (Active Comparator): Standard ablation power parameters (40-45 W)
  Interventions: Procedure: Standard ablation power

INTERVENTIONS:
Procedure: High power ablation — High power ablation parameters (50-55 W)
  Arms: High power ablation
Procedure: Standard ablation power — Standard ablation power parameters (40-45 W)
  Arms: Standard ablation power

SUMMARY:
Background: Patient's freedom from VT after RFA remains non-optimal and it depends on many factors. One of them is the effective reduction of the myocardium with RF energy during the operation. The standardization of the parameters of RF will help to increase the success of the procedure.

Hypothesis: Radiofrequency ablation of ventricular tachycardias with high power parameters has comparable safety and leads to greater efficacy (absence of ventricular tachycardias and all types of cardioverter-defibrillator therapies) in the long-term compared with ablation with standard parameters in patients with structural heart disease.

Purpose: to evaluate the safety and the efficiency of ablation of ventricular tachycardia in patients with structural heart disease using high power RF energy.

DETAILED DESCRIPTION:
Background: Patient's freedom from VT after RFA remains non-optimal and it depends on many factors. One of them is the effective reduction of the myocardium with RF energy during the operation. The standardization of the parameters of RF will help to increase the success of the procedure.

Hypothesis: Radiofrequency ablation of ventricular tachycardias with high power parameters has comparable safety and leads to greater efficacy (absence of ventricular tachycardias and all types of cardioverter-defibrillator therapies) in the long-term compared with ablation with standard parameters in patients with structural heart disease.

Purpose: to evaluate the safety and the efficiency of ablation of ventricular tachycardia in patients with structural heart disease using high power RF energy.

Tasks:

1. To analyze the number of intraoperative complications in both groups
2. To evaluate the number of recurrent ventricular tachycardias and the number of episodes of CDI therapy in the long-term follow-up period
3. To estimate the time of onset of the first episode of VT and the overall burden of VT in the long-term follow-up period
4. To compare the total time of surgery, fluoroscopy, the number and total time of RF exposure, as well as the ablation index in relation to the "acute" and separated efficiency of ablation in the study groups
5. To estimate all-cause mortality in both groups
6. The number of repeated ablation for recurrent VT
7. The number of justified and unfounded CDI therapies
8. To analyze the long-term burden of antiarrhythmic therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients after myocardial infarction (at least 3 months before enrollment in the study)
2. Stable, documented, monomorphic VT, confirmed by ECG and / or CMECG and / or EGM of any implanted device, having appropriate rhythm discrimination algorithms
3. Patients who have signed the informed consent

Exclusion Criteria:

1. Acute myocardial ischemia
2. A reversible cause of VT (e.g. drug arrhythmia), recently(up to 30 days) suffered from acute coronary syndrome, coronary revascularization (<90 days for bypass surgery, <30 days for percutaneous coronary intervention), or having functional class IV angina.
3. Thrombosis of the left ventricle
4. Patients who have been implanted the mechanical prostheses in the aortic and mitral positions.
5. Patients who have been performed the catheter RFA for VT.
6. Renal failure (creatinine clearance <15 ml / min),
7. Patients with NYHA functional class IV heart failure
8. Patients with a medical condition that may limit survival to less than 1 year
9. Patients with myocardial infarction with ST-segment elevation or MI without ST-segment elevation, transferred less than 30 days ago.
10. Patients who haven't signed the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
The number of intraoperative complications | Day 1
  The number of intraoperative complications (death, hemopericardium, stroke, heart attack, electrical storm, vascular complications)
The inducibility of the clinical VT at the end of ablation procedure | Day 1
  The number of patients with inducible VT at the end of the ablation procedure
The number of recurrent ventricular tachycardias | Up to one year
  The number of recurrent ventricular tachycardias on one-year follow-up period after single procedure
The number of episodes of ICD therapy | Up to one year
  The number of episodes of ICD therapy on one-year follow-up period after single procedure

SECONDARY OUTCOMES:
Freedom from recurrent VT | 3 months
  Time to the first episode of VT on 3 months follow-up period after single procedure
The total time of ablation procedure | Up to one year
  The total time of ablation procedure
The total time of fluoroscopy | Up to one year
  The total time of fluoroscopy
The total number of RF exposures | Up to one year
  The total number of RF exposures
The total time of RF exposures | Up to one year
  The total time of RF exposures
All-cause mortality | Up to one year
  All-cause mortality (Time to any death occurring at any time on one-year follow-up period )
The number of redo ablation procedures for recurrent VT | Up to one year
  The number of redo ablation procedures for recurrent VT on one-year follow-up period
The number of appropriate and unappropriated ICD therapies | Up to one year
  The number of appropriate and unappropriated ICD therapies
The number of antiarrhythmic drugs | Up to one year
  The number of antiarrhythmic drugs on one-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V. Korolev, MD, Principal Investigator — Federal Research Clinical Center FMBA Russia
Locations (7):
- Texas Cardiac Arrhythmia Institute, Austin, Texas, United States
- Heart and Vascular Center, Bad Bevensen, Germany
- Russia (5):
  - Federal Research Clinical Center of Federal Medical & Biological Agency, Moscow
  - National Medical Research Center of Surgery named after A. Vishnevsky, Moscow
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - National Medical Research Center of Cardiology, Moscow
  - Meshalkin National Medical Research Center, Novosibirsk

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data (IPD).